CLINICAL TRIAL: NCT04780022
Title: Patent Foramen Ovale Closure in Older Patients: A Collaborative Multicenter Retrospective Study
Brief Title: Patent Foramen Ovale Closure in Older Patients
Acronym: PFO-Elderly
Status: Completed | Type: Observational
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Collaborators: Toronto General Hospital (Other); Montreal Heart Institute (Other); Ottawa Heart Institute (Unknown); St. Boniface Hospital (Other); Hospital Clinico de Madrid (Unknown); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Other Study IDs: PFO-Elderly
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Patent Foramen Ovale; Ischemic Stroke; Older People
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older patients with cryptogenic embolism and PFO closure: Data (clinical events at last follow-up) on patients older than 60 years who have experienced a previous paradoxical embolism of unknown origin and underwent transcatheter PFO closure will be collected.
  Interventions: Other: Clinical events at last follow-up

INTERVENTIONS:
Other: Clinical events at last follow-up — Clinical events (stroke, transient ischemic attack, peripheral embolism, deep venous thrombosis, atrial fibrillation, myocardial infarction, bleeding episode, death) at last follow-up

SUMMARY:
* Describe the baseline and procedural characteristics of older patients undergoing PFO closure due to cryptogenic embolism.
* Assess the long-term follow-up of this cohort, focusing on neurological events and their origin, major cardiac outcomes, as well as survival rates and death origin.
* Seek for predictors of neurological event recurrence after the procedure.

DETAILED DESCRIPTION:
In patients with cryptogenic stroke, up to 4 randomized trials and subsequent meta-analyses have recently shown a significant reduction in recurrent ischemic stroke events following percutaneous closure of patent foramen ovale (PFO) . All randomized trials but one excluded patients older than 60 years, and a mean patient age of about 50 years was reported in the single randomized trial including older patients. Thus, whereas PFO closure has been established as the new gold-standard therapy in young patients with cryptogenic stroke and PFO, there are no definite recommendations on the management of patients older than 60 years. Some studies have shown that older patients with cryptogenic stroke exhibit a much higher prevalence of PFO (compared with patients with stroke of known cause), similar to that in younger populations, but scarce data exist on acute and mid-term clinical outcomes of older patients undergoing PFO closure.

The investigators have recently reported the results of study comparing the long-term clinical outcomes of patients older (vs. younger) than 60 years in our centre. A total of 475 consecutive patients (90 older than 60 years) were included, and the main results can be summarized as follows: 1) older patients with cryptogenic embolism and PFO exhibited a higher burden of cardiovascular risk factors; 2) PFO closure was safe in older patients, with no differences in periprocedural complications compared with younger patients; 3) at long-term (median of 8 years) follow-up post-PFO closure, the global mortality rate was higher among older patients, but differences were driven by noncardiovascular mortality (mainly cancer), and 4) the rate of recurrent stroke/TIA was low (much lower than that predicted by the RoPE score), but there was a tendency toward a higher incidence of recurrent stroke/TIA among older patients, which appeared to be partially related to cardiovascular risk factor burden (no differences in recurrent ischemic event rate were observed after adjustment for baseline differences in cardiovascular risk factors between groups). The main limitation of this study was the relatively low number of patients older than 60 years, precluding an appropriate evaluation of the factors associated with poorer clinical outcomes in this population. Thus, the investigators are planning to confirm prior findings in a collaborative project including a much larger cohort of patients. Also, the results of this retrospective study would provide the rationale for a CIHR submission on a randomized trial targeting this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years who have experienced a previous paradoxical embolism (stroke, transient ischaemic attack or peripheral embolism) of unknown origin and underwent transcatheter PFO closure.

Exclusion Criteria:

* PFO closure indication other than paradoxical embolism (example: platypnea orthodeoxia syndrome).
* Surgical PFO closure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 60 years who have experienced a previous paradoxical embolism of unknown origin and underwent transcatheter PFO closure.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of stroke | Through study completion, an average of 1 year
Rate of transient ischemic attack | Through study completion, an average of 1 year
Rate of peripheral embolism | Through study completion, an average of 1 year
Rate of deep venous thrombosis | Through study completion, an average of 1 year
Rate of atrial fibrillation | Through study completion, an average of 1 year
Rate of myocardial infarction | Through study completion, an average of 1 year
Rate of bleeding | Through study completion, an average of 1 year
Rate of death | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUCPQ, Québec, Quebec, Canada

REFERENCES:
- [Background] Sondergaard L, Kasner SE, Rhodes JF, Andersen G, Iversen HK, Nielsen-Kudsk JE, Settergren M, Sjostrand C, Roine RO, Hildick-Smith D, Spence JD, Thomassen L; Gore REDUCE Clinical Study Investigators. Patent Foramen Ovale Closure or Antiplatelet Therapy for Cryptogenic Stroke. N Engl J Med. 2017 Sep 14;377(11):1033-1042. doi: 10.1056/NEJMoa1707404. PMID 28902580
- [Background] Mas JL, Derumeaux G, Guillon B, Massardier E, Hosseini H, Mechtouff L, Arquizan C, Bejot Y, Vuillier F, Detante O, Guidoux C, Canaple S, Vaduva C, Dequatre-Ponchelle N, Sibon I, Garnier P, Ferrier A, Timsit S, Robinet-Borgomano E, Sablot D, Lacour JC, Zuber M, Favrole P, Pinel JF, Apoil M, Reiner P, Lefebvre C, Guerin P, Piot C, Rossi R, Dubois-Rande JL, Eicher JC, Meneveau N, Lusson JR, Bertrand B, Schleich JM, Godart F, Thambo JB, Leborgne L, Michel P, Pierard L, Turc G, Barthelet M, Charles-Nelson A, Weimar C, Moulin T, Juliard JM, Chatellier G; CLOSE Investigators. Patent Foramen Ovale Closure or Anticoagulation vs. Antiplatelets after Stroke. N Engl J Med. 2017 Sep 14;377(11):1011-1021. doi: 10.1056/NEJMoa1705915. PMID 28902593
- [Background] Saver JL, Carroll JD, Thaler DE, Smalling RW, MacDonald LA, Marks DS, Tirschwell DL; RESPECT Investigators. Long-Term Outcomes of Patent Foramen Ovale Closure or Medical Therapy after Stroke. N Engl J Med. 2017 Sep 14;377(11):1022-1032. doi: 10.1056/NEJMoa1610057. PMID 28902590
- [Background] Lee PH, Song JK, Kim JS, Heo R, Lee S, Kim DH, Song JM, Kang DH, Kwon SU, Kang DW, Lee D, Kwon HS, Yun SC, Sun BJ, Park JH, Lee JH, Jeong HS, Song HJ, Kim J, Park SJ. Cryptogenic Stroke and High-Risk Patent Foramen Ovale: The DEFENSE-PFO Trial. J Am Coll Cardiol. 2018 May 22;71(20):2335-2342. doi: 10.1016/j.jacc.2018.02.046. Epub 2018 Mar 12. PMID 29544871
- [Background] Wintzer-Wehekind J, Alperi A, Houde C, Cote JM, Del Val D, Cote M, Rodes-Cabau J. Transcatheter closure of patent foramen ovale in patients older than 60 years of age with cryptogenic embolism. Rev Esp Cardiol (Engl Ed). 2020 Mar;73(3):219-224. doi: 10.1016/j.rec.2019.07.003. Epub 2019 Oct 1. English, Spanish. PMID 31585849
- [Background] Kent DM, Ruthazer R, Weimar C, Mas JL, Serena J, Homma S, Di Angelantonio E, Di Tullio MR, Lutz JS, Elkind MS, Griffith J, Jaigobin C, Mattle HP, Michel P, Mono ML, Nedeltchev K, Papetti F, Thaler DE. An index to identify stroke-related vs incidental patent foramen ovale in cryptogenic stroke. Neurology. 2013 Aug 13;81(7):619-25. doi: 10.1212/WNL.0b013e3182a08d59. Epub 2013 Jul 17. PMID 23864310